CLINICAL TRIAL: NCT03203291
Title: The Integration of Motor Learning Principles to Reduce Load Asymmetry Using a Novel Robotic Device in Individuals Chronically Post-Stroke
Brief Title: Reducing Asymmetry During Gait Using the TPAD (Tethered Pelvic Assist Device) for Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Sunil Agrawal, Professor of Mechanical Engineering and of Rehabilitation and Regenerative Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAR2407
Record Dates: First submitted 2017-06-24; First posted 2017-06-29 (Actual); Results first posted 2019-10-28 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Stroke
Keywords: stroke; robotic training; gait
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Tethered Pelvic Assist Device (TPAD) Treatment (Experimental): All participants will receive 5 consecutive days of training with the TPAD (tethered pelvic assist device) with testing completed before training, on completion of training and at a 1-week follow up.
  Interventions: Device: TPAD (Tethered Pelvic Assist Device)

INTERVENTIONS:
Device: TPAD (Tethered Pelvic Assist Device) — Each day of intervention will include a 1-hour treadmill based intervention to promote increased loading onto the affected limb. Visual feedback will be provided and faded over the course of the 5-day training. Immediately on completion of the treadmill intervention, participants will receive an additional 5-10 minutes of overground intervention reinforcing weight shifting onto the affected limb.

SUMMARY:
OBJECTIVES: The purpose of this study is to evaluate the overall feasibility in terms of safety, treatment tolerance and adherence as well as preliminarily address how effective this treatment model using the TPAD and overground training would be to reduce load asymmetry on the treadmill and promote increased stance symmetry on the paretic limb during overground gait.PARTICIPANTS: A total of 12 individuals in the chronic (>6 months) stages post stroke will be recruited from a voluntary stroke research database for participation. DESIGN: A non-randomized pilot study of feasibility will be used to establish the feasibility and preliminary efficacy of using the TPAD in combination with overground training to reduce load force asymmetry in this population. METHODS: Participants will undergo a series of three assessments within a one-week time frame prior to initiating intervention. Intervention using the TPAD and overground training will occur during week 2 over 5 consecutive visits (Mon-Fri). Participants will also complete short walks before and after the intervention with an instrumented system that records individual walking characteristics. Participants will return one-week after completing the intervention for a final test of walking and balance. Each study visit will be approximately 1-1.5 hours in duration, and total participation should be completed within three weeks. EXPECTED OUTCOMES: We anticipate this training paradigm will prove feasible and effective in reducing both load and stance asymmetry in a population of individuals with chronic stroke.

DETAILED DESCRIPTION:
There are a number of common impairments resulting from stroke that contribute to motor deficits which affect gait, or walking ability. These manifest as decreased walking speed, and further, as stroke affects only one side of the body, there are resulting asymmetries in time, spatial and force parameters during walking. Robotic-based therapies have been used to increase walking speed and reduce asymmetry in a population of individuals after stroke, however these therapies have demonstrated results similar to that of non-robotic, or conventional training. This is possibly due to the control strategies used in robotic training, which strategies limit participant involvement and reduce learning effect. The Tethered Pelvic Assist Device (TPAD) is a robotic device that uses motorized tethers attached to a belt at the user's pelvis to guide the pelvis along a pre-set movement trajectory. These tethers can be configured in an infinite array of possibilities, and most recently have been used to facilitate a body weight shift onto the paretic limb in a population of individuals after stroke. Other robotic devices constrain the limb through the entire movement trajectory and constrict the participants ability to participate in motor planning and movement execution. The TPAD promotes weight shifting, but allows an individual to freely move the limb and to navigate leg movement and foot placement independently, without constraints. Further, if coupled with overground training to promote transfer of improvements to walking over ground, this device maybe useful at improving symmetry in individuals after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (>6 months) post stroke
* Single stroke event
* Montreal Cognitive Assessment (MoCA) score of >22
* Independently ambulating in the home
* Use of a unilateral assistive device (e.g. cane)
* Marked asymmetry in stance phase (defined by a symmetry ratio < 0.90)

Exclusion Criteria:

* History of multiple strokes
* History of other neurological disease
* Uncontrolled medical issues
* Muscle contractures of the lower limb limiting range of motion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Agrawal, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bishop L, Omofuma I, Stein J, Agrawal S, Quinn L. Treadmill-Based Locomotor Training With Robotic Pelvic Assist and Visual Feedback: A Feasibility Study. J Neurol Phys Ther. 2020 Jul;44(3):205-213. doi: 10.1097/NPT.0000000000000317. PMID 32516301

RESULTS

PARTICIPANT FLOW:
Groups:
- TPAD Treatment: All participants will receive 5 consecutive days of training with the TPAD (tethered pelvic assist device) with testing completed before training, on completion of training and at a 1-week follow up.
  TPAD (Tethered Pelvic Assist Device): Each day of intervention will include a 1-hour treadmill based intervention to promote increased loading onto the affected limb. Visual feedback will be provided and faded over the course of the 5-day training. Immediately on completion of the treadmill intervention, participants will receive an additional 5-10 minutes of overground intervention reinforcing weight shifting onto the affected limb.
Period: Overall Study
Arm/Group | TPAD Treatment
Started | 12
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | TPAD Treatment
Number analyzed (Participants) | 11
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 50.18 (11.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11
Months Since Stroke [Mean (Standard Deviation); unit: months] | 71.24 (46.70)

OUTCOME MEASURES:

1. Primary Outcome: Force Symmetry Ratio During Gait
Description: 0-1 symmetry ratio comparing the impulse force of the affected limb versus the unaffected limb during gait. If the unaffected limb performs equivalent to the affected limb, the ratio has a value of 1. The greater the disparity between limbs, the closer the ratio is to 0.
Time Frame: Baseline through day 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | TPAD Treatment
Number analyzed (Participants) | 11
ratio
  Baseline | 0.71 (0.09)
  Day 5 | 0.83 (0.23)

2. Primary Outcome: Stance Time Symmetry Ratio
Description: 0-1 symmetry ratio of the percentage of time spent in the stance phase of a gait cycle. If the unaffected limb performs equivalent to the affected limb, the ratio will have a value of 1. The greater the disparity the closer the ratio is to 0.
  Stance time symmetry = Time in stance phase of gait cycle of Affected/Unaffected limb.
Time Frame: Baseline through week 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | TPAD Treatment
Number analyzed (Participants) | 11
ratio
  Baseline | 0.81 (0.04)
  Day 5 | 0.86 (0.05)
  Week 3 | 0.83 (0.05)

3. Secondary Outcome: Symmetry Ratio of Stride Length
Description: 0-1 symmetry ratio comparing the stride length of the affected limb versus the unaffected limb during gait. If the unaffected limb performs equivalent to the affected limb, the ratio has a value of 1. The greater the disparity between limbs, the closer the ratio is to 0.
Time Frame: Baseline through week 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | TPAD Treatment
Number analyzed (Participants) | 11
ratio
  Baseline | 1.04 (0.05)
  Day 5 | 1.06 (0.08)
  Week 3 | 1.03 (0.05)

4. Secondary Outcome: Gait Velocity
Description: Walking velocity (speed) measured in meters walked per second (measured by Inertial Measurement Unit sensors worn in real time during walking).
Time Frame: Baseline through week 3
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | TPAD Treatment
Number analyzed (Participants) | 11
meters/second
  Baseline | 0.56 (0.22)
  Day 5 | 0.57 (0.20)
  Week 3 | 0.59 (0.25)

5. Secondary Outcome: Symmetry of Percentage of Time in Swing Phase of Gait
Description: 0-1 symmetry ratio compares the amount of time the unaffected leg is in swing phase of the gait cycle compared to the affected leg. The swing phase means the period of time during the gait cycle when one foot is not in contact with the ground. If the unaffected limb performs equivalent to the affected limb, the ratio has a value of 1. The greater the disparity between limbs, the closer the ratio is to 0.
Time Frame: Baseline through week 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | TPAD Treatment
Number analyzed (Participants) | 11
ratio
  Baseline | 0.66 (0.11)
  Day 5 | 0.73 (0.11)
  Week 3 | 0.68 (0.12)

6. Secondary Outcome: Time Spent in Double Support Phase of Gait
Description: The percentage of time in one gait cycle spent in double support phase of gait (2 feet in contact with the ground).
Time Frame: Baseline through week 3
Measure: Mean (Standard Deviation); unit: percentage of gait cycle
Arm/Group | TPAD Treatment
Number analyzed (Participants) | 11
percentage of gait cycle
  Baseline | 31.62 (9.74)
  Day 5 | 34.12 (8.53)
  Week 3 | 31.76 (10.38)

7. Secondary Outcome: Berg Balance Scale
Description: Berg Balance Scale measures balance ability of adults. The scale has 14 items, each is rated on a 5-point scale ranging from 0-4. A score of 0 indicates the lowest level of function and 4 indicating the highest level of function. Total scores range from 0-56, with higher scores indicating better balance.
Time Frame: Baseline through week 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TPAD Treatment
Number analyzed (Participants) | 11
units on a scale
  Baseline | 48.00 (5.45)
  Day 5 | 49.09 (4.72)
  Week 3 | 49.18 (4.69)

ADVERSE EVENTS:
Time Frame: Baseline through week 3.
Arm/Group | TPAD Treatment
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT03203291/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT03203291/SAP_001.pdf